CLINICAL TRIAL: NCT01776931
Title: Determination of Lysine Requirements in Healthy Pregnant Women Using the Indicator Amino Acid Oxidation Technique
Brief Title: Determination of Lysine Requirements in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H11-02435
Record Dates: First submitted 2013-01-17; First posted 2013-01-28 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Pregnancy
Keywords: Indicator Amino acid technique; Lysine requirements; Pregnancy; Dietary protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lysine intake (Experimental): Dietary supplement:lysine intake
  Interventions: Dietary Supplement: Lysine intake

INTERVENTIONS:
Dietary Supplement: Lysine intake — Oral consumption of Eight hourly experimental meals- Includes 4 tracer-free experimental meals containing a mixture of free amino acids, calories from a flavored liquid and protein free cookies and 4- labeled amino acid experimental meals.

SUMMARY:
Amino acids are building blocks of protein in our body. It is important that pregnant women eat adequate amount of protein/amino acids to ensure healthy growth and development of the fetus.Lysine is an amino acid that is present in high amounts only in animal foods (meat) and not much in plant foods such as wheat. Currently , it is not known how much lysine is needed to eat during pregnancy.

Current Dietary Reference Intake recommendations for amino acid requirements are based on non-pregnant adults, and minimally based on pregnancy-specific data.To the investigators knowledge, there is no scientific information regarding the amount of lysine needed at different stages of pregnancy.

The investigators hypothesize that current recommendations for lysine intake in pregnant women are underestimated. The investigators also hypothesize that the lysine requirements will be greater during the later stages of pregnancy, compared to early stages.

The purpose of this study is to determine lysine requirements in healthy pregnant women 19-40y,(1st and 3rd trimester) using a modern, safe and quick technique called the indicator amino acid oxidation technique and to compare lysine requirements during early (15-18 weeks last menstrual period) late (33-36 weeks last menstrual period) stages of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Maternal age 19-40y
* Early stage of pregnancy(15-18 weeks) and late stage of pregnancy(33-36 weeks)
* In good health (free of chronic/acute illness, full range of physical mobility)
* Healthy pre-pregnancy body mass index

Exclusion Criteria:

* Subjects outside the age range of 19-40y
* Women pregnant with more than one child
* Body mass Index less than 18.5kg/m2 or greater than 25 kg/m2
* less than 18 months between current pregnancy and last pregnancy
* History of spontaneous abortion,pre-term birth, preeclampsia/eclampsia, gestational diabetes, pregnancy-related anemia, pregnancy related jaundice
* Existing metabolic disease
* Substance dependance (i.e. alcohol, cigarette, illicit drugs)
* Allergic to eggs and egg protein
* Severe nausea and vomiting during pregnancy

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
13 carbon dioxide production | 8 hours (1 study day)
  Urine and breath samples will be collected during the study to measure the rate of oxidation of tracer in expired breath and flux by enrichment in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — Child & Family Research Institute/University of British Columbia
Locations (1):
- Child & Family Research Institute, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Payne M, Stephens T, Lim K, Ball RO, Pencharz PB, Elango R. Lysine Requirements of Healthy Pregnant Women are Higher During Late Stages of Gestation Compared to Early Gestation. J Nutr. 2018 Jan 1;148(1):94-99. doi: 10.1093/jn/nxx034. PMID 29378056